CLINICAL TRIAL: NCT02903979
Title: Impact of Different Restorative Treatments for Deep Caries Lesion in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Ibirapuera (Other)
Responsible Party: Principal Investigator, Tamara Kerber Tedesco, PhD in Pediatric Dentistry, Universidade Ibirapuera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIB1
Record Dates: First submitted 2016-09-06; First posted 2016-09-16 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Deep Caries Lesion of Primary Teeth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- HVGIC (Experimental): Restorations with only HVGIC in deep caries lesion of primary teeth.
  Interventions: Other: HVGIC
- Indirect pulp capping (Active Comparator): Indirect pulp capping with calcium hydroxide cement, restored with HVGIC:
  Interventions: Other: Indirect pulp capping

INTERVENTIONS:
Other: HVGIC — In experimental group, the researches will be performed a restoration, after partial caries removal, with high viscosity glass ionomer cement in the teeth with deep caries lesion.
  Arms: HVGIC
Other: Indirect pulp capping — In control group, the researches will be performed a indirect pulp capping with calcium hydroxide cement and high viscosity glass ionomer cement in the teeth with deep caries lesion.
  Arms: Indirect pulp capping

SUMMARY:
In front of a lack of evidence to determine the best treatment for deep cavitated carious lesions, the search for an effective restorative technique, which results in a least possible discomfort to patients, and reduce the time needed for the restorative treatment, if becomes relevant. The objective of this randomized clinical trial to evaluate the efficacy of high viscosity glass ionomer cement restorations (HVGIC) compared to restoration with calcium hydroxide restoration associated with high viscosity glass ionomer cement (HVGIC) for treatment of deep lesions in primary molars, as well as the impact of treatment in the criteria focused on the patient as well as cost-efficacy of the techniques . Children with 4 to 8 years will be selected randomly at the Clinic for Children at the University Ibirapuera of Dentistry. 108 teeth will be randomized into two groups: (1) restoration with calcium hydroxide cement associated with HVGIC and (2) HVGIC restoration. The restorations will be evaluated after 6, 12 and 24 months by two trained examiners blinded to the treatments. The efficacy of each treatment is measured by four main outcomes, which are: (1) criteria related to the effectiveness of the restorative treatment (2) criteria focused on the patient and (3) cost-efficacy. For comparison between the two groups will be used the Kaplan-Meier survival and the long-rank test. Cox regression is performed the assessment of the influence of some other variable results. For all analyzes, the significance level is set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included that have at least one primary molar with deep cavitated carious lesions in occlusal surface.

Exclusion Criteria:

* Patients will be excluded with special needs, using orthodontics devices and / or systemic diseases which may affect the oral cavity. Also, teeth with pulp exposure, spontaneous pain, mobility, presence of abscess or fistula next to the tooth, teeth with restorations, sealants or enamel formation defects will also be excluded.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Pulp Vitality | Up to 24 months
  To evaluate the survival of different restorative treatments considering the pulp vitality.

SECONDARY OUTCOMES:
Wong-Baker scale to discomfort | Immediately to restoration procedure.
  To evaluate the discomfort of different restorative treatments by a Wong-Baker scale.
Cost-efficacy analysis by total value of treatment in relation to efficacy | Up to 24 months
  To evaluate the cost-efficacy of different restorative treatments by total value in dollar of treatment in relation to efficacy. The researchers would like to analyze that a treatment of low cost show the similar efficacy of a high cost treatment.
Restoration longevity | Up to 24 months.
  To evaluate the restoration longevity by clinical examination.
Caries progression | Up to 24 months.
  To evaluate the caries progression by radiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Ibirapuera, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] da Silva GSQ, Raggio DP, Machado GFR, Mello-Moura ACV, Gimenez T, Floriano I, Tedesco TK. Impact of different restorative treatments for deep caries lesion in primary teeth (CEPECO 1) - study protocol for a noninferiority randomized clinical trial. BMC Oral Health. 2019 Jan 8;19(1):6. doi: 10.1186/s12903-018-0703-3. PMID 30621659